CLINICAL TRIAL: NCT01378481
Title: High-Dose Vorinostat With Radiation Therapy in the Treatment of Recurrent Glioma
Brief Title: High-Dose Vorinostat and Fractionated Stereotactic Body Radiation Therapy in Treating Patients With Recurrent Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01139; NCI-2012-01139 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11D.101 (Other: Thomas Jefferson University Hospital); 9018 (Other: CTEP); P30CA056036 (NIH)
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-03

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Mixed Glioma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma; Brain Neoplasms | interventions — Vorinostat; Radiosurgery

ARMS (1):
- Treatment (vorinostat, surgery, FSRT) (Experimental): Patients receive high-dose vorinostat PO at 48, 27, and 3 hours prior to surgery. Beginning 2-6 weeks later, patients receive vorinostat PO QD on days 1-3 in weeks 1-2and undergo fractionated stereotactic body radiation therapy on days 1-5 in weeks 1-2. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Vorinostat; Radiation: Stereotactic Radiosurgery; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Vorinostat — Given PO
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid
Radiation: Stereotactic Radiosurgery — Undergo fractionated stereotactic radiation therapy
  Other Names: SBRT; Stereotactic External Beam Irradiation; Stereotactic Radiation Therapy; Stereotactic Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Procedure: Therapeutic Conventional Surgery — Undergo neurosurgery

SUMMARY:
This study is being done to determine if an investigational cancer treatment called vorinostat combined with fractionated stereotactic radiation therapy (FSRT) is effective in treating recurrent high grade gliomas. The main goal of this research study is to determine the highest dose of vorinostat that can be given to patients with recurrent tumors. The study will also determine the potential side effects and safety of these treatment combinations. Vorinostat is a small molecule inhibitor of histone deacetylase (HDAC). HDAC inhibitors help unravel the deoxyribonucleic acid (DNA) of the cancer cells and make them more susceptible to the treatment with radiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the phase II dose when intermittent short-course vorinostat is combined with fractionated radiation therapy in recurrent high-grade glioma.

SECONDARY OBJECTIVES:

I. Define the pharmacokinetics of vorinostat entry into the cerebrospinal fluid (CSF) and demonstrate that vorinostat influences glioma biology.

OUTLINE: This is a dose-escalation study of vorinostat.

Patients receive high-dose vorinostat orally (PO) at 48, 27, and 3 hours prior to surgery. Beginning 2-6 weeks later, patients receive vorinostat PO once daily (QD) on days 1-3 in weeks 1-2and undergo fractionated stereotactic body radiation therapy on days 1-5 in weeks 1-2. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a previously histologically or cytologically confirmed glioma (astrocytic or oligodendroglial supratentorial tumors grades 3 or 4 according to the World Health Organization [WHO] 2007 classification) that has been previously treated with fractionated radiation therapy and now shows evidence of recurrence
* Patients must have recovered from the toxic effects of prior therapy
* Patients must have recovered from the effects of any prior surgery to any part of the body; there must be a minimum of 28 days from the day of surgery to the day of registration; for core or needle biopsy, a minimum of 7 days must have elapsed prior to registration
* Patients may have previously undergone more than one craniotomy
* Prior treatment with cytotoxic and biological agents is permissible; there should be at least a 2 week break between prior treatment and enrollment; (in the case of bevacizumab, since this trial involves surgery, at least 4 weeks should elapse between last dose of drug and enrollment, in the case of nitrosoureas or mitomycin C, at least 6 weeks)
* Prior treatment with fractionated radiation therapy (up to 60 Gray [Gy]) is an eligibility criterion, however this should have been completed >= 4 weeks prior to enrollment and there should not have been a second course of fractionated radiotherapy to the supratentorial area
* One prior single fraction radiosurgical procedure within the treatment field is acceptable if V12 < 5 cc (V12 is the volume of brain receiving 12 or more Gy); additional radiosurgical procedures outside of the treatment area are acceptable
* Patients should not have received prior histone deacetylase therapy (HDAC) therapy, an exception being the anti-seizure medicine valproic acid; however even valproic acid should not be given concurrently with vorinostat
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 2 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Prothrombin time/international normalized ratio (PT INR) < 1.4 for patients not on warfarin
* Women of childbearing potential must have a negative beta-human chorionic gonadotropin (HCG) pregnancy test documented within 7 days prior to registration
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; the effects of vorinostat on the developing human fetus are unknown; HDAC inhibitor agents as well as the ionizing radiation used in this trial are known to be teratogenic; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had:

  * Radiotherapy within 4 weeks
  * Chemotherapy/biological agents (excluding bevacizumab, nitrosoureas and mitomycin C) within 2 weeks
  * Bevacizumab within 4 weeks
  * Nitrosoureas and mitomycin C within 6 weeks prior to entering the study
  * Those who have not recovered from acute adverse events due to any prior therapeutic agents
* Patients may not be receiving any other investigational agents
* Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an electrocardiogram (EKG) performed within 14 days of registration
* A history of long QT syndrome, or corrected QTc (QTc) prolongations > 470 ms at baseline
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or other HDAC inhibitor or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because vorinostat is an antineoplastic agent with the potential for teratogenic or abortifacient effects, class D; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, breastfeeding should be discontinued if the mother is treated with vorinostat; these potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD), defined as one level below at which 2 of 6 patients experience a dose-limiting toxicity (DLT) | 48 hours
  Analysis of study data will be descriptive, including summary tables of toxicity. An exploratory retrospective trend analysis will be performed assessing for a correlation between plasma drug level and toxicity, using exact logistic regression models.
Dose limiting toxicities (grade 3 or higher) defined by Common Toxicity Criteria (CTC) version 4.0 | 48 hours
  Analysis of study data will be descriptive, including summary tables of toxicity. An exploratory retrospective trend analysis will be performed assessing for a correlation between plasma drug level and toxicity, using exact logistic regression models.
Overall survival (OS) | Up to 2 years
  Analysis of study data will be descriptive, including Kaplan-Meier estimates of survival outcomes.
Progression free survival (PFS) | Time from start of treatment to time to progression, up to 2 years
  Analysis of study data will be descriptive, including Kaplan-Meier estimates of survival outcomes.
Response rate defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Up to 2 years
  Analysis of study data will be descriptive. A 2-sided exact 95% confidence interval of response rate will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States